CLINICAL TRIAL: NCT00102557
Title: Hydroxychloroquine Versus Clobetasol 0.05% Rinse for the Treatment of Oral Lichen Planus
Brief Title: Hydroxychloroquine vs. Clobetasol Rinse to Treat Oral Lichen Planus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050086; 05-D-0086
Record Dates: First submitted 2005-01-29; First posted 2005-01-31 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-10

CONDITIONS: Lichen Planus, Oral
Keywords: Vesiculobullous; Mucosal Lesions; Oral Health; Dermatology; Plaquenil; Oral Lichen Planus; Mouth Lesions; Oral Lesions
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine

SUMMARY:
This study will compare two treatments for oral lichen planus - hydroxychloroquine (Plaquenil) tablets and clobetasol oral rinse. Oral lichen planus is a chronic disorder in which patients have painful mouth ulcers that interfere with meals and daily functioning. It is most commonly treated with topical or systemic corticosteroids, but these drugs have a number of side effects, most commonly yeast infection, and chronic systemic use of them can lead to diabetes, osteoporosis, weight gain, and other complications. Also, lichen planus generally returns when the corticosteroids are stopped. Clobetasol oral rinse is a topical steroid commonly used to treat oral lichen planus. Hydroxychloroquine, a drug that was originally used to treat malaria and is now also approved for lupus and rheumatoid arthritis, has been tried for lichen planus in small-scale studies with some evidence of benefit.

Patients 18 years of age and older with oral lichen planus may be eligible for this study. Pregnant women are excluded. Candidates are screened with a dermatology examination, routine blood tests, an eye examination, and a biopsy to rule out other conditions similar to lichen planus and to provide tissue for research purposes. For the biopsy, two small circles of tissue about 4 mm (less than 1/5") across are surgically removed from the area with lichen planus.

Participants are randomly assigned to treatment with either hydroxychloroquine or clobetasol rinse. Patients assigned to hydroxychloroquine also take a placebo mouth rinse that looks and tastes like the clobetasol rinse, and those assigned to clobetasol also take a pill that looks and tastes like the hydroxychloroquine tablet. This is done so that neither the patients nor the study doctors know which patient is taking which active medication until the study is completed. Patients take the pills daily in the morning with food or a glass of milk for the 6-month study period and use the rinse twice a day for 4 months and then once a day for 2 months. They may not use any pain or anti-inflammatory medicines or topical creams, gels or rinses regularly, because these medications can obscure the effects of the study drugs and complicate interpretation of the results. They are given a topical numbing medicine as part of the study and can use Tylenol for pain during the study duration.

In addition to treatment, participants visit the NIH Clinical Center once a month for the following tests and procedures:

* Review of pain levels, as recorded in a pain diary
* Review of drug side effects, if any
* Collection of saliva and blood samples at 2, 4 and 6 months
* Repeat oral biopsy at completion of the study at 6 months to evaluate treatment effects
* Final examination at 8 months to determine if the disease returns or improves after the medication is stopped.

DETAILED DESCRIPTION:
This is a randomized double blind parallel group trial of safety and efficacy of hydroxychloroquine in oral lichen planus and associated cutaneous and genital lesions.

The primary objective of the study is to test the hypothesis that oral hydroxychloroquine taken at 6mg/kg of lean weight will be at least as effective as clobetasol rinse in healing ulcerations associated with the erosive form of lichen planus. Secondary objectives will include assessment of changes in salivary and tissue proteome and plasma, saliva, and tissue cytokine profiles over the course of treatment with hydroxychloroquine and clobetasol. We hope that this will allow us to gain insight in the pathophysiology of mucosal lichen planus as well as the mechanism of action of hydroxychloroquine in this condition.

Total surface area of oral erosions will be the primary outcome in this study. We will consider 50% reduction in ulcerated area over 6 months clinically significant. Secondary outcomes will include changes in two lichen planus severity scales, reduction of pain levels as measured by a visual analogue scale and amount of topical analgesic used, improvement in oral and systemic disease-specific and generic quality of life scores. We will also assay plasma, saliva, and tissue cytokines over the course of the study to assess dynamics of cytokine levels in this disease. We will evaluate salivary proteome changes associated with disease activity using 2D gel electrophoresis and mass spectrometric methods.

The principal study interventions will be hydroxychloroquine at 6 mg/kg of lean weight or clobetasol 0.05% oral rinse. Additional allowed interventions will be standard oral topical analgesic rinse on an as needed basis. Diagnostic and research evaluations will include ophthalmologic screening prior to enrollment and at the completion of the study, complete history and oral and general physical examination, laboratory investigations, saliva collection, and oral mucosal biopsy at the start and finish of the study. The total period of time that each subject will spend in the interventional period of the trial will be 6 months. Additional off study follow-up period will be 2 months.

ELIGIBILITY:
INCLUSION CRITERIA:

Biopsy confirmed symptomatic erosive oral lichen planus. World Health Organization histological criteria (21) in combination with compatible clinical picture will be used for diagnosis. In questionable cases, direct immunofluorescence will be performed to exclude other conditions.

No current treatment with hydroxychloroquine or other immunomodulatory agents. A one-month washout period will be required prior to enrollment if patients are taking immunomodulatory agents. Prior treatment with topical steroids will be allowed.

Age greater than 18 years old. Lichen planus is very rare in patients younger than 40 years old and children are especially sensitive to the effects of hydroxychloroquine.

Patients of both sexes and all racial and ethnic groups will be eligible.

The presence of at least one ulcerated oral lesion with a surface area of at least 100 sq. mm as measured bi-directionally.

EXCLUSION CRITERIA:

Unable to undergo oral biopsy for diagnosis

Lichen planus with no ulcerated oral lesions of greater than 100 sq. mm in area.

Treatment with hydroxychloroquine or other immunomodulatory agents within 1 month of the randomization.

Hepatitis B or Hepatitis C infection

Significant abnormalities in hepatic status as measured by liver function tests (ALT, AST, AP, bilirubin.) Mild asymptomatic elevations in liver enzymes (up to 20% above the reference range) will not preclude enrollment in the trial.

Significant abnormalities in renal status as measured by kidney function tests (creatinine, BUN).

Uncontrolled diabetes

Contraindications to hydroxychloroquine or clobetasol therapy (known hypersensitivity, retinopathy from prior use, history of aplastic anemia or agranulocytosis).

Anemia (defined as a hemoglobin level more than 2 standard deviations below the mean reference value for age).

Granulocytopenia (defined as an absolute neutrophil count (ANC) in adults as less than 1500/mm(3)).

Pregnancy or lactation. Pregnancy status will be assessed by questionnaire. Potentially pregnant patients will be evaluated by plasma HCG test. Patients planning pregnancy will be excluded. Sexually active females will be required to use contraception prior to enrollment in the study. Every woman of childbearing age will have a pregnancy test.

Inability or unwillingness to give written informed consent.

Serious concurrent disease (e.g. myocardial infarction, severe heart failure, severe COPD) requiring hospitalization or limiting life expectancy to less than 1 year.

Psoriasis

G6PD deficiency

Porphyria

Chronic use of non-steroidal anti-inflammatory agents or other agents to relieve pain.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74
Dates: Start 2005-01; Study Completion 2005-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Dental And Craniofacial Research (NIDCR), Bethesda, Maryland, United States

REFERENCES:
- [Background] Axell T, Rundquist L. Oral lichen planus--a demographic study. Community Dent Oral Epidemiol. 1987 Feb;15(1):52-6. doi: 10.1111/j.1600-0528.1987.tb00480.x. PMID 3467894
- [Background] Eisen D. The clinical manifestations and treatment of oral lichen planus. Dermatol Clin. 2003 Jan;21(1):79-89. doi: 10.1016/s0733-8635(02)00067-0. PMID 12622270
- [Background] Scully C, Beyli M, Ferreiro MC, Ficarra G, Gill Y, Griffiths M, Holmstrup P, Mutlu S, Porter S, Wray D. Update on oral lichen planus: etiopathogenesis and management. Crit Rev Oral Biol Med. 1998;9(1):86-122. doi: 10.1177/10454411980090010501. PMID 9488249